CLINICAL TRIAL: NCT01182675
Title: Hematopoietic Stem Cell Transplantation for Children With Severe Combined Immunodeficiency Disease Utilizing Alemtuzumab and Mobilization With Plerixafor & Filgrastim
Brief Title: Hematopoietic Stem Cell Transplantation (HSCT) for Children With SCID Utilizing Alemtuzumab, Plerixafor & Filgrastim
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient evidence of efficacy
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Christopher Dvorak, Assistant Professor, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSF10-00701
Record Dates: First submitted 2010-08-09; First posted 2010-08-17 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Severe Combined Immunodeficiency
Keywords: SCID; Transplant; Alemtuzumab; Plerixafor
MeSH Terms: conditions — Severe Combined Immunodeficiency | interventions — Transplantation Conditioning; Filgrastim; plerixafor; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-cell Graft Permissive SCID (Experimental): Patients with SCID with:
  i. NK- phenotype; ii. NK+ phenotype with 10/10 HLA-matched relative or unrelated donor; or iii. NK+ phenotype with maternal engraftment by STR analysis and undergoing haplocompatible HSCT from maternal donor Intervention: Transplant Conditioning with Mobilization Only
  Interventions: Drug: Transplant Conditioning with Mobilization Only
- T-cell Graft Resistant SCID (Experimental): Patients with SCID with NK+ phenotype with HLA-mismatched donor Intervention: Transplant Conditioning with Mobilization and Alemtuzumab
  Interventions: Drug: Transplant Conditioning with Mobilization and Alemtuzumab

INTERVENTIONS:
Drug: Transplant Conditioning with Mobilization Only — Day -4: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -3: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -2: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -1: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day 0: Plerixafor 240 mcg/kg subcutaneous 9-12 hours prior to transplant; Day 0 Transplant
  Other Names: Conditioning with Filgrastim and Plerixafor
  Arms: T-cell Graft Permissive SCID
Drug: Transplant Conditioning with Mobilization and Alemtuzumab — Day -7: Alemtuzumab 0.3 mg test dose then 0.3 mg/kg IV; Day -6: Alemtuzumab 0.3 mg/kg IV; Day -5: Alemtuzumab 0.3 mg/kg IV; Day -4: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -3: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -2: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -1: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day 0: Plerixafor 240 mcg/kg subcutaneous 9-12 hours prior to transplant; Day 0: Transplant
  Other Names: Conditioning with Filgrastim, Plerixafor, and Alemtuzumab
  Arms: T-cell Graft Resistant SCID

SUMMARY:
The goal of this study is to develop a novel approach to hematopoietic stem cell transplantation for children with Severe Combined Immunodeficiency Disease (SCID) that eliminates the use of toxic chemotherapy conditioning and maximizes the likelihood of T and B cell immune reconstitution. Rather than classic chemotherapeutic agents, the investigators will utilize a targeted stem cell mobilizer, plerixafor, in combination with alemtuzumab, a monoclonal antibody. Correlative scientific questions will include: 1) efficacy and characteristics of host stem cell mobilization; and 2) alemtuzumab pharmacokinetics in very young children.

DETAILED DESCRIPTION:
The goal of this study is to develop an approach to hematopoietic stem cell transplantation for children with Severe Combined Immunodeficiency Disease (SCID) that eliminates the use of toxic chemotherapy conditioning and maximizes the likelihood of T and B cell immune reconstitution. SCID is a rare primary immunodeficiency disease in which there are multiple genotypes and phenotypes, and depending on various factors including the presence of B cell and NK cells, and the presence of maternal cells in the patient's circulation, there are numerous ways to approach a transplant. The major issues that must be addressed in any approach to transplantation for SCID are graft rejection and T and B cell immune reconstitution. Depending on the specific SCID diagnosis, the phenotype, and the presence of maternal engraftment at diagnosis, we will evaluate two transplant approaches that will attempt to optimize the engraftment of donor HSC and the likelihood of T and B cell reconstitution while eliminating the use of toxic chemotherapy conditioning.

1. Primary Objective: To determine if the administration of plerixafor & filgrastim (G-CSF) prior to stem cell infusion results in increased donor stem cell occupancy of available bone marrow niches and B-cell engraftment in patients with SCID.
2. Secondary Objectives:

i. To determine if NK cell depletion with Alemtuzumab will overcome NK-mediated graft resistance in haplocompatible transplants for NK+ SCID.

ii. To determine the optimal dosing of Alemtuzumab in very young children. iii. To determine the immunophenotypic characteristics of CD34+ cells mobilized and engrafted in patients receiving plerixafor & filgrastim prior to HCT.

iv. To determine the thymic output, as measured by T-cell receptor excision circles, in patients receiving haplocompatible transplants & boosts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with classic SCID phenotype (<400 CD3/ul or maternally engrafted and <10% of normal PHA lymphoproliferative response). Genotypic identification is preferable, but not required.
* Patients must have an acceptable stem cell donor (HLA matched relative, 9 or 10/10 HLA-matched unrelated, or haplocompatible relative).

Exclusion Criteria:

* Patients with "leaky" SCID syndromes, Omenn's Syndrome, reticular dysgenesis, ADA deficiency
* Lansky score <60%
* Patient with expected survival <4 weeks (including disseminated CMV infection involving lungs and/or CNS)

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2010-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Dvorak, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Dvorak CC, Hung GY, Horn B, Dunn E, Oon CY, Cowan MJ. Megadose CD34(+) cell grafts improve recovery of T cell engraftment but not B cell immunity in patients with severe combined immunodeficiency disease undergoing haplocompatible nonmyeloablative transplantation. Biol Blood Marrow Transplant. 2008 Oct;14(10):1125-1133. doi: 10.1016/j.bbmt.2008.07.008. PMID 18804042
- [Background] Dvorak CC, Cowan MJ. Radiosensitive severe combined immunodeficiency disease. Immunol Allergy Clin North Am. 2010 Feb;30(1):125-42. doi: 10.1016/j.iac.2009.10.004. PMID 20113890
- [Background] Dvorak CC, Cowan MJ. Hematopoietic stem cell transplantation for primary immunodeficiency disease. Bone Marrow Transplant. 2008 Jan;41(2):119-26. doi: 10.1038/sj.bmt.1705890. Epub 2007 Oct 29. PMID 17968328

RESULTS

PARTICIPANT FLOW:
Groups:
- T-cell Graft Permissive SCID: Patients with SCID with:
  i. NK- phenotype; ii. NK+ phenotype with 10/10 HLA-matched relative or unrelated donor; or iii. NK+ phenotype with maternal engraftment by STR analysis and undergoing haplocompatible HSCT from maternal donor
  Transplant Conditioning with Mobilization Only: Day -4: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -3: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -2: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -1: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day 0: Plerixafor 240 mcg/kg subcutaneous 9-12 hours prior to transplant; Day 0 Transplant
- T-cell Graft Resistant SCID: Patients with SCID with NK+ phenotype with HLA-mismatched donor
  Transplant Conditioning with Mobilization and Alemtuzumab: Day -7: Alemtuzumab 0.3 mg test dose then 0.3 mg/kg IV; Day -6: Alemtuzumab 0.3 mg/kg IV; Day -5: Alemtuzumab 0.3 mg/kg IV; Day -4: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -3: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -2: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -1: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day 0: Plerixafor 240 mcg/kg subcutaneous 9-12 hours prior to transplant; Day 0: Transplant
Period: Overall Study
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID
Started | 7 | 0
Completed | 7 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients with T-cell Graft Resistant SCID were enrolled during the time the trial was open.
Groups:
- Total: Total of all reporting groups
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID | Total
Number analyzed (Participants) | 7 | 0 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 |  | 7
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Engraftment of Donor B-cells in Blood by STR Testing
Description: Number of participants in whom donor B cells were detected in the patient's blood after HSCT.
Time Frame: 1 Year
Population: No patients with T-cell Graft Resistant SCID were enrolled during the time the trial was open.
Measure: Number; unit: participants
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID
Number analyzed (Participants) | 7 | 0
participants | 0 |

2. Secondary Outcome: Incidence of Acute GVHD
Time Frame: 100 Days
Population: No patients with T-cell Graft Resistant SCID were enrolled during the time the trial was open.
Measure: Number; unit: participants
Groups:
- T-cell Graft Permissive SCID: Patients with SCID with:
  i. NK- phenotype; ii. NK+ phenotype with 10/10 HLA-matched relative or unrelated donor; or iii. NK+ phenotype with maternal engraftment by STR analysis and undergoing haplocompatible HSCT from maternal donor Intervention: Transplant Conditioning with Mobilization Only
  Transplant Conditioning with Mobilization Only: Day -4: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -3: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -2: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day -1: Filgrastim (G-CSF) 5 mcg/kg IV q12 hours; Day 0: Plerixafor 240 mcg/kg subcutaneous 9-12 hours prior to transplant; Day 0 Transplant
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID
Number analyzed (Participants) | 7 | 0
participants | 1 |

3. Secondary Outcome: Incidence of Chronic GVHD
Time Frame: 2 Years
Population: No patients with T-cell Graft Resistant SCID were enrolled during the time the trial was open.
Measure: Count of Participants; unit: Participants
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID
Number analyzed (Participants) | 7 | 0
Participants | 1 |

4. Secondary Outcome: Percentage of Patients Who Become Independent From Regular IVIG Infusion
Description: Based on B-cell function assays from the patient's blood, we will be able to determine if patients are able to successfully discontinue IVIG infusions.
Time Frame: 2 Years
Population: No patients with T-cell Graft Resistant SCID were enrolled during the time the trial was open.
Measure: Count of Participants; unit: Participants
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID
Number analyzed (Participants) | 7 | 0
Participants | 0 |

5. Secondary Outcome: Number of Patients With Engraftment of Donor Stem Cells in Bone Marrow by STR Testing
Description: We will measure whether we are able to detect donor stem cells in the patient's bone marrow after HSCT.
Time Frame: 1 Year
Population: No patients with T-cell Graft Resistant SCID were enrolled during the time the trial was open.
Measure: Count of Participants; unit: Participants
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID
Number analyzed (Participants) | 7 | 0
Participants | 0 |

6. Secondary Outcome: Number of Patients Who Achieve Engraftment of Donor T-cells in Blood by STR Testing
Description: We will measure whether we are able to detect donor T-cells in the patient's blood after HSCT.
Time Frame: 1 Year
Population: No patients with T-cell Graft Resistant SCID were enrolled during the time the trial was open.
Measure: Count of Participants; unit: Participants
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID
Number analyzed (Participants) | 7 | 0
Participants | 7 |

ADVERSE EVENTS:
Description: No patients with T-cell Graft Resistant SCID were enrolled during the time the trial was open.
Arm/Group | T-cell Graft Permissive SCID | T-cell Graft Resistant SCID
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/0
Other Adverse Events (participants affected / at risk) | 0/7 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No